CLINICAL TRIAL: NCT00114036
Title: Trial to Reduce Antimicrobial Prophylaxis Errors (TRAPE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: Joint Commission on Accreditation of Healthcare Organizations (Other); Society for Healthcare Epidemiology of America (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R01HS011331-01A1 (AHRQ)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Cardiovascular Surgical Procedures; Arthroplasty, Replacement; Hysterectomy
Keywords: Antibiotic prophylaxis; Surgical wound infections
MeSH Terms: conditions — Surgical Wound Infection

INTERVENTIONS:
Behavioral: Quality improvement strategies

SUMMARY:
The specific aims are to determine the incidence of medication errors related to antimicrobial prophylaxis for cardiovascular surgery, joint replacement surgery, and hysterectomies across a heterogeneous sample of hospitals; identify organizational and practitioner factors associated with error rates, and evaluate the effectiveness of a multifaceted intervention in reducing prophylaxis error rates compared to written feedback alone in a sample of 44 hospitals enrolled in the study using a rigorous group-randomized design.

DETAILED DESCRIPTION:
Numerous studies have shown that many surgical site infections (SSI) are preventable with appropriately timed antimicrobial prophylaxis. Patients receiving prophylaxis either well-before or well after surgery are up to 5 times more likely to develop an SSI than those receiving appropriate therapy (Classen et al, 1992). Unfortunately, errors in antimicrobial prophylaxis timing are extremely common with error rates typically reported to be between 35 and 40%. Given that errors in antimicrobial prophylaxis are common and the consequences of error so grave, identifying methods to assist hospitals in improving prophylaxis must be a high priority. TRAPE will evaluate a multifaceted, theory-based intervention to assist hospitals in progressing through stages of organizational change to improve the prophylaxis process. We will test the impact of the intervention using a rigorous group-randomized, nested, pretest-posttest design (Murray, 1998).

Our specific aims over the 4 year project period are:

1. determine the incidence of medication errors related to antimicrobial prophylaxis for cardiovascular surgery, joint replacement surgery, and hysterectomies in 44 hospitals recruited to participate in the study;
2. identify organizational and system factors associated with error rates;
3. randomize the 44 hospitals to evaluate the effectiveness of a multifaceted intervention.

The interventions consist of: a) the promotion of specific process changes likely to reduce error rates, b) a site-visit, c) customized process feedback, d) facilitated benchmarking, and e) peer consultation. The 22 intervention hospitals will be compared to 22 hospitals that receive written feedback of their error rates only. The study has 80% power to detect a 12-15% improvement in the timing of prophylaxis in the full intervention group compared to the written feedback only group. Data collection will be done at each participating hospital, and the medical records of 100 surgical patients before and after the intervention will be abstracted at each hospital to establish performance rates. Changes in the processes of care, and the evolution through stages of organizational change will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals with a minimum number of surgeries per month

Age Groups: Child, Adult, Older Adult
Dates: Start 2002-08; Study Completion 2005-12

PRIMARY OUTCOMES:
Change in performance between hospitals in the intervention and hospitals in the control group on the proportion of prophylaxis administered within the recommended timeframes.

SECONDARY OUTCOMES:
Change in performance on appropriate selection of drug, appropriate duration, appropriate number of doses pre-op, appropriate use of beta-lactams in patients with allergies.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Krichevsky, PhD, Principal Investigator — Wake Forest University Health Sciences; Barbara I. Braun, PhD, Study Director — Joint Commission on Accreditation of Healthcare Organizations; Edward Wong, MD, Study Chair — VA Office of Research and Development; Steve Solomon, MD, Study Chair — Centers for Disease Control and Prevention; Bryan Simmons, MD, Study Chair — Methodist Health System; Andrew J. Bush, PhD, Study Chair — University of Tennessee; John Burke, MD, Study Chair — LDS Hospital; Michele R. Bozikis, MPH, Study Chair — Joint Commission on Accreditation of Healthcare Organizations; Linda Kusek, MPH, Study Chair — Joint Commission on Accreditation of Healthcare Organizations
Locations (3):
- United States (3):
  - Joint Commission on Accreditation of Healthcare Organizations, Oakbrook Terrace, Illinois
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Derived] Kritchevsky SB, Braun BI, Bush AJ, Bozikis MR, Kusek L, Burke JP, Wong ES, Jernigan J, Davis CC, Simmons B; TRAPE Study Group. The effect of a quality improvement collaborative to improve antimicrobial prophylaxis in surgical patients: a randomized trial. Ann Intern Med. 2008 Oct 7;149(7):472-80, W89-93. doi: 10.7326/0003-4819-149-7-200810070-00007. PMID 18838727